CLINICAL TRIAL: NCT05044975
Title: Improving Sleep in Gynecologic Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rina Fox, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00213356; K08CA247973 (NIH)
Record Dates: First submitted 2021-09-03; First posted 2021-09-16 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-02

CONDITIONS: Sleep Disturbance; Gynecologic Cancer
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Sleep restriction, Stimulus control, and Systematic light exposure (Experimental)
  Interventions: Behavioral: Sleep restriction; Behavioral: Stimulus control; Behavioral: Systematic light exposure
- Sleep restriction and Stimulus control (Experimental)
  Interventions: Behavioral: Sleep restriction; Behavioral: Stimulus control
- Sleep restriction and Systematic light exposure (Experimental)
  Interventions: Behavioral: Sleep restriction; Behavioral: Systematic light exposure
- Stimulus control and Systematic light exposure (Experimental)
  Interventions: Behavioral: Stimulus control; Behavioral: Systematic light exposure
- Sleep Restriction (Experimental)
  Interventions: Behavioral: Sleep restriction
- Stimulus control (Experimental)
  Interventions: Behavioral: Stimulus control
- Systematic light exposure (Experimental)
  Interventions: Behavioral: Systematic light exposure
- Sleep tracking (No Intervention)

INTERVENTIONS:
Behavioral: Sleep restriction — Participants will receive sleep restriction intervention
  Arms: Sleep Restriction; Sleep restriction and Stimulus control; Sleep restriction and Systematic light exposure; Sleep restriction, Stimulus control, and Systematic light exposure
Behavioral: Stimulus control — Participants will receive stimulus control intervention
  Arms: Sleep restriction and Stimulus control; Sleep restriction, Stimulus control, and Systematic light exposure; Stimulus control; Stimulus control and Systematic light exposure
Behavioral: Systematic light exposure — Participants will receive systematic light exposure intervention
  Arms: Sleep restriction and Systematic light exposure; Sleep restriction, Stimulus control, and Systematic light exposure; Stimulus control and Systematic light exposure; Systematic light exposure

SUMMARY:
This purpose of this study is to learn about how to provide treatment to gynecologic cancer survivors who have difficulty sleeping.

DETAILED DESCRIPTION:
This study has two parts.

In Part 1, 15 gynecologic cancer survivors will receive three candidate intervention components known to reduce sleep disturbance (i.e., sleep restriction, stimulus control, systematic light exposure) simultaneously for six weeks. Participants will then complete semi-structured individual interviews to provide feedback about barriers to and facilitators of intervention adherence. Results of Part 1 will inform the design and delivery of the candidate components in Part 2.

In Part 2, a 2^3 full factorial design will be followed to randomize 80 gynecologic cancer survivors to one of eight six-week intervention conditions reflecting all possible combinations of the three candidate intervention components.

ELIGIBILITY:
Inclusion Criteria:

* History of Stage I, II, or III gynecologic cancer
* Age 18+ years
* English language proficiency
* Current sleep disturbance demonstrated by a Pittsburgh Sleep Quality Index (PSQI) score > 5
* Usual sleep onset time between 9:00PM and 3:00AM
* Reliable telephone and Internet access

Exclusion Criteria:

* Stage IV disease
* Diagnosed or suspected psychiatric or medical condition that may interfere with participation (e.g., psychosis, dementia, bipolar disorder, abuse of alcohol or illicit substances within the past 6 months, narrow angle glaucoma, retinal disorders, epilepsy or a similar condition)
* Diagnosed sleep apnea, narcolepsy, periodic limb movement disorder, or restless legs syndrome unless well controlled
* Use of medications that may be contraindications for study procedures due to safety concerns or due to potential impact on intervention efficacy or assessment validity (e.g., sedatives/hypnotics), to be identified on a case-by-case basis
* Shift worker
* Severe physical or cognitive impairment (≥ 2 errors on a brief six-item version of the Mini Mental State Exam [MMSE] or Patient Reported Functional Status [PRFS] score > 2, which is based on the Eastern Cooperative Oncology Group [ECOG]but has been modified to be in lay language)
* Plans to travel across 3 or more meridians/time zones during the 6 intervention weeks or plans to cross any meridians/time zones during the 2 weeks leading up to wearing an actiwatch.
* History of a primary diagnosis of a distinct non-gynecologic or non-skin cancer other than a non-melanoma skin cancer within the 5 years prior to enrollment
* For participants with Stage III ovarian cancer: less than 2 years post-completion of primary gynecologic cancer treatment and/or less than 60 days post-surgery. For patients with any other gynecologic cancer/stage: less than 30 days post-completion of primary gynecologic cancer treatment and/or less than 60 days post-surgical intervention (e.g., hysterectomy)
* Male
* Have received CBT-I or systematic bright light therapy within the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in objectively-measured sleep outcomes from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Wrist actigraphy
Changes in subjectively-reported sleep quality from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Subjectively-reported sleep quality over the past 7 days will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance questionnaire. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the underlying construct.
Changes in perceived impairment during wake associated with sleep problems from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Perceived impairment during wake associated with sleep problems over the past seven days will be measured with the PROMIS Sleep-Related Impairment questionnaire. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the underlying construct.

SECONDARY OUTCOMES:
Changes in health-related quality of life (HRQOL) from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  The 27-item Functional Assessment of Cancer Therapy - General (FACT-G) will measure HRQOL.
Changes in overall symptom burden from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  The 32-item Memorial Symptom Assessment Scale (MSAS) will evaluate symptom burden.
Changes in symptoms of depression from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Symptoms of depression over the past seven days with be measured with the PROMIS Depression questionnaire. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the underlying construct.
Changes in symptoms of anxiety from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Symptoms of anxiety over the past seven days with be measured with the PROMIS Anxiety questionnaire. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the underlying construct.
Changes in fatigue from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Fatigue over the past seven days with be measured with the PROMIS Fatigue questionnaire. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the underlying construct.

OTHER OUTCOMES:
Changes in circadian activity rhythms from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  Wrist actigraphy
Changes in urinary 6-Sulfatoxymelatonin from baseline to immediately after the intervention and 3-months post-intervention | Baseline (Part 1 and Part 2 participants), immediately after the intervention (Part 1 and Part 2 participants), 3-months post-intervention (Part 2 participants only)
  The night prior to each assessment participants will collect overnight urine to enable analysis of urinary 6-Sulfatoxymelatonin

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona College of Nursing, Tucson, Arizona
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox RS, Gaumond JS, Zee PC, Kaiser K, Tanner EJ, Ancoli-Israel S, Siddique J, Penedo FJ, Wu LM, Reid KJ, Parthasarathy S, Badger TA, Rini C, Ong JC. Optimizing a Behavioral Sleep Intervention for Gynecologic Cancer Survivors: Study Design and Protocol. Front Neurosci. 2022 Mar 4;16:818718. doi: 10.3389/fnins.2022.818718. eCollection 2022. PMID 35310101